CLINICAL TRIAL: NCT02614066
Title: A Phase 1/2 Multi-Center Study Evaluating the Safety and Efficacy of KTE-X19 in Adult Subjects With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (r/r ALL) (ZUMA-3)
Brief Title: A Study Evaluating the Safety and Efficacy of Brexucabtagene Autoleucel (KTE-X19) in Adult Subjects With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (ZUMA-3)
Acronym: ZUMA-3
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTE-C19-103; 2015-005009-35 (EudraCT Number)
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2021-11-29 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Recurrence | interventions — brexucabtagene autoleucel; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: 2 x 10^6 Anti-CD19 CAR T Cells/kg (Experimental): Participants with relapsed or refractory B-precursor acute lymphoblastic leukemia (r/r B-ALL) will receive conditioning chemotherapy (fludarabine 25 mg/m^2 intravenously [IV] over 30 minutes on Day -4, Day -3, and Day -2 and cyclophosphamide 900 mg/m^2 IV over 60 minutes on Day -2) following a single IV infusion of brexucabtagene autoleucel (KTE-X19) chimeric antigen receptor (CAR) transduced autologous T cells at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of body weight on Day 0. For participants weighing > 100 kg, a maximum flat dose of 2 x 10^8 anti-CD19 CAR T cells/kg of body weight will be administered.
  Interventions: Biological: brexucabtagene autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Phase 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg (Experimental): Participants with r/r B-ALL will receive conditioning chemotherapy (fludarabine 25 mg/m^2 IV over 30 minutes on Day -4, Day -3, and Day -2 and cyclophosphamide 900 mg/m^2 IV over 60 minutes on Day -2) following a single IV infusion of brexucabtagene autoleucel CAR transduced autologous T cells at a target dose of 1 x 10^6 anti-CD19 CAR T cells/kg of body weight on Day 0. For participants weighing > 100 kg, a maximum flat dose of 1 x 10^8 anti-CD19 CAR T cells/kg of body weight will be administered.
  Interventions: Biological: brexucabtagene autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Phase 1: 0.5 x 10^6 Anti-CD19 CAR T Cells/kg (Experimental): Participants with r/r B-ALL will receive conditioning chemotherapy (fludarabine 25 mg/m^2 IV over 30 minutes on Day -4, Day -3, and Day -2 and cyclophosphamide 900 mg/m^2 IV over 60 minutes on Day -2) following a single IV infusion of brexucabtagene autoleucel CAR transduced autologous T cells at a target dose of 0.5 x 10^6 anti-CD19 CAR T cells/kg of body weight on Day 0. For participants weighing > 100 kg, a maximum flat dose of 0.5 x 10^8 anti-CD19 CAR T cells/kg of body weight will be administered.
  Interventions: Biological: brexucabtagene autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg (Experimental): Participants with r/r B-ALL will receive conditioning chemotherapy (fludarabine 25 mg/m^2 IV over 30 minutes on Day -4, Day -3, and Day -2 and cyclophosphamide 900 mg/m^2 IV over 60 minutes on Day -2) following a single IV infusion of brexucabtagene autoleucel CAR transduced autologous T cells at a target dose of 1 x 10^6 anti-CD19 CAR T cells/kg of body weight on Day 0. For participants weighing > 100 kg, a maximum flat dose of 1 x 10^8 anti-CD19 CAR T cells/kg of body weight will be administered.
  Interventions: Biological: brexucabtagene autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: brexucabtagene autoleucel — A single infusion of brexucabtagene autoleucel CAR transduced autologous T cells administered intravenously.
  Other Names: KTE-X19
Drug: Cyclophosphamide — Administered intravenously.
Drug: Fludarabine — Administered intravenously.

SUMMARY:
The primary objectives of this study are to determine the safety and efficacy of brexucabtagene autoleucel (KTE-X19) in adult participants with relapsed/refractory (r/r) B-precursor acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
Bridging therapy could be administered at the discretion of the investigator and is recommended for participants with high disease burden at baseline (M3 marrow [> 25% leukemic blasts] or ≥ 1,000 blasts/mm^3 in the peripheral circulation) to control participant's disease prior to conditioning chemotherapy. Bridging therapy includes:

Attenuated VAD: Vincristine non-liposomal (1-2 mg IV weekly) or liposomal (2.25 mg/m^2 IV weekly), and dexamethasone 20-40 mg IV or oral administration (PO) daily x 3-4 days per week. Optional doxorubicin 50 mg/m^2 IV x 1 (first week only).

Mercaptopurine (6-MP): 50-75 mg/m^2/day by mouth (administer at bedtime on an empty stomach to improve absorption).

Hydroxyurea: Doses titrated between 15-50 mg/kg/day (rounded to the nearest 500 mg capsule and given as a single daily oral dose on a continuous basis).

DOMP: Dexamethasone 6 mg/m^2/day PO (or IV) divided twice daily (BID) Days 1-5, vincristine 1.5 mg/m^2 (maximum dose 2 mg) IV on Day 1, methotrexate 20 mg/m^2 PO weekly, 6-MP 50- 75mg/m^2/day PO daily.

Attenuated FLAG/FLAG-IDA: fludarabine 30 mg/m^2 IV days 1-2, cytarabine 2 g/m^2 IV days 1-2, G-CSF 5 μg/kg subcutaneously (SC) or IV starts on Day 3 and can continue until day before the start of conditioning chemotherapy. With or without idarubicin 6 mg/m^2 IV Days 1-2.

Mini-hyper CVAD (courses A and/or B):

* Course A: Cyclophosphamide 150 mg/m^2 every 12 hours x 3 days, dexamethasone 20 mg/d IV or PO daily Days 1-4 and 11-14, vincristine 2 mg IV x 1
* Course B: Methotrexate 250 mg/m^2 IV over 24 hours on Day 1,cytarabine 0.5 g/m^2 IV every 12 hours x 4 doses on Days 2 and 3.

After completion of the Month 24 visit, subjects who received an infusion of KTE-X19 will complete the remainder of the 15 year follow-up assessments in a separate long-term follow-up study, KT-US-982-5968

ELIGIBILITY:
Key Inclusion Criteria:

1. Relapsed or refractory B-precursor ALL defined as one of the following:

   * Primary refractory disease
   * First relapse if first remission ≤ 12 months
   * Relapsed or refractory disease after 2 or more lines of systemic therapy
   * Relapsed or refractory disease after allogeneic transplant provided individuals is at least 100 days from stem cell transplant at the time of enrollment
2. Morphological disease in the bone marrow (≥ 5% blasts)
3. Individuals with Philadelphia chromosome positive (Ph+) disease are eligible if they are intolerant to tyrosine kinase inhibitor (TKI) therapy, or if they have relapsed/refractory disease despite treatment with at least 2 different TKIs
4. Eastern cooperative oncology group (ECOG) performance status of 0 or 1
5. Adequate renal, hepatic, pulmonary and cardiac function defined as:

   * Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 cc/min
   * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN)
   * Total bilirubin ≤ 1.5 mg/dl, except in individuals with Gilbert's syndrome.
   * Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion, and no clinically significant arrhythmias
   * Baseline oxygen saturation > 92% on room air
6. In individuals previously treated with blinatumomab, cluster of differentiation 19 (CD19) tumor expression in bone marrow or peripheral blood.

Key Exclusion Criteria:

1. Diagnosis of Burkitt's leukemia/lymphoma according to World Health Organization (WHO) classification or chronic myelogenous leukemia lymphoid blast crisis
2. History of malignancy other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease free for at least 3 years
3. Isolated extramedullary disease
4. Central nervous system (CNS) abnormalities

   * Presence of CNS-3 disease or CNS-2 disease with neurological changes
   * History or presence of any CNS disorder such as a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
5. History of concomitant genetic syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman-Diamond syndrome or any other known bone marrow failure syndrome
6. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment
7. History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment.
8. Primary immunodeficiency
9. Known infection with human immunodeficiency virus (HIV), hepatitis B (HBsAg positive) or hepatitis C virus.
10. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management.
11. Prior medication:

    * Salvage chemotherapy including TKIs for Ph+ ALL within 1 week prior to enrollment
    * Prior CD19 directed therapy other than blinatumomab
    * Treatment with alemtuzumab within 6 months prior to leukapheresis, or treatment with clofarabine or cladribine within 3 months prior to leukapheresis
    * Donor lymphocyte infusion (DLI) within 28 days prior to enrollment
    * Any drug used for graft-versus-host disease (GVHD) within 4 weeks prior to enrollment
    * At least 3 half-lives must have elapsed from any prior systemic inhibitory/stimulatory immune checkpoint molecule therapy prior to enrollment
    * Corticosteroid therapy for 7 days prior to enrollment
12. Presence of any indwelling line or drain (e.g., percutaneous nephrostomy tube, indwelling Foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter). Ommaya reservoirs and dedicated central venous access catheters such as a Port-a-Cath or Hickman catheter are permitted
13. Acute GVHD grade II-IV by Glucksberg criteria or severity B-D by International Bone Marrow Transplant Registry (IBMTR) index; acute or chronic GVHD requiring systemic treatment within 4 weeks prior to enrollment
14. Live vaccine ≤ 4 weeks prior to enrollment
15. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential
16. Individuals of both genders of child-bearing potential who are not willing to practice birth control from the time of consent through 6 months after the completion of brexucabtagene autoleucel (KTE-X19)
17. In the investigators judgment, the individuals is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation
18. History of autoimmune disease (e.g. Crohns, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2022-07-23 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (33):
- United States (22):
  - UC San Diego-Moores Cancer Center, La Jolla, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Loyola University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of MD Greenbaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Tisch Cancer Institute, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, New York, New York
  - Sarah Cannon, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Center, Seattle, Washington
- University Health Network - Princess Margaret, Toronto, Ontario, Canada
- France (4):
  - Institut Paoli Calmettes, Marseille
  - Hopital Saint Louis, Paris
  - Hopital Haut-Leveque, Pessac
  - Hopital Pontchaillou - CHU de Rennes - Service d'Hematologie, Rennes
- Germany (3):
  - Universitatsklinikum Frankfurt, Frankfurt
  - Klinikum der Universitat Munchen, München
  - Universitaetsklinikum Wuerzburg, Würzburg
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Result] Oluwole OO, Shah BD, Baer MR, Bishop MR, Holmes H, Schiller GJ, et al. Outcomes of Patients with Relapsed/Refractory Acute Lymphoblastic Leukemia Treated with Prior Blinatumomab in ZUMA-3, a Study of KTE-C19, an Anti-CD19 Chimeric Antigen Receptor (CAR) T Cell Therapy [Abstract S1569]. The 23rd European Hematology Association (EHA) Congress 2018 14-17 June; Stockholm, Sweden.
- [Result] Sabatino M, Choi K, Chiruvolu V, Better M. Production of Anti-CD19 CAR T Cells for ZUMA-3 and -4: Phase 1/2 Multicenter Studies Evaluating KTE-C19 in Patients With Relapsed/Refractory B-Precursor Acute Lymphoblastic Leukemia (R/R ALL) [Abstract 711]. Blood 2016;128 (22):1227.
- [Result] Shah B, Castro J, Gokbuget N, Kersten MJ, Hagenbeek T, Wierda W, et al. ZUMA-3: A Phase 1/2 Multi-center Study Evaluating the Safety and Efficacy of KTE-C19 Anti-CD19 CAR T Cells in Adult Subjects with Relapsed/Refractory B Precursor Acute Lymphoblastic Leukemia (r/r ALL). European Society for Medical Oncology (ESMO) Congress 2016;Abstract 3713.
- [Result] Shah B, Huynh V, Sender LS, Lee DW, Castro JE, Wierda WG, et al. High Rates of Minimal Residual Disease-Negative (MRD-) Complete Responses (CR) in Adult and Pediatric and Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia (R/R ALL) Treated With KTE-C19 (Anti-CD19 Chimeric Antigen Receptor [CAR] T Cells): Preliminary Results of the ZUMA-3 and ZUMA-4 Trials. Blood 2016;128 (22):2803.
- [Result] Shah B, Stock W, Wierda W, Topp M, Kersten MJ, Houot R, et al. KTE-C19, an Anti-CD19 Chimeric Antigen Receptor (CAR) T cell Therapy in Adult Patients (Pts) With Relapsed/ Refractory Acute Lymphoblastic Leukemia (R/R ALL) in the ZUMA-3 Trial: Preliminary Results of Novel Safety Interventions [Abstract ALL-025]. Clinical lymphoma, myeloma & leukemia 2017;17:S253.
- [Result] Shah B, Stock W, Wierda W, Topp MS, Kersten MJ, Houot R, et al. Preliminary Results of Novel Safety Interventions in Adult Patients (Pts) With Relapsed/Refractory Acute Lymphoblastic Leukemia (R/R ALL) in the ZUMA-3 Trial. European Society for Medical Oncology (ESMO) Congress 2017.
- [Result] Shah B, Wierda WG, Schiller GJ, Bishop MR, Castro JE, Sabatino M, et al. KTE-C19 Chimeric Antigen Receptor (CAR) T Cell Therapy in Adults with High-Burden Relapsed/Refractory Acute Lymphoblastic Leukemia (R/R ALL): Updated Results from Phase 1/2 of ZUMA-3 [Abstract P523]. The 22nd European Hematology Association (EHA) Congress 2017 22-25 June; Madrid, Spain.
- [Result] Shah BD, Bishop MR, Oluwole OO, Logan A, Baer MR, Donnellan WB, et al. End of Phase I Results of ZUMA-3, A Phase 1/2 Study of KTE-X19, Anti-CD19 Chimeric Antigen Receptor (CAR) T Cell Therapy, in Adult Patients (pts) with Relapsed/Refractory (R/R) Acute Lymphoblastic Leukemia (ALL) [Abstract]. J Clin Oncol 2019;37 (15):7006.
- [Result] Shah BD, Bishop MR, Oluwole OO, Logan AC, Baer MR, Donnellan WB, et al. KTE-X19, an Anti-CD19 Chimeric Antigen Receptor T Cell Therapy, in Adult Patients with Relapsed/Refractory Acute Lymphoblastic Leukemia: End of Phase 1 Results of ZUMA-3 [Abstract PS945]. HemaSphere 2019;3 (S1):426.
- [Result] Shah BD, Oluwole OO, Baer MR, Bishop MR, Holmes H, Schiller GJ, et al. KTE-C19, an Anti-CD19 Chimeric Antigen Receptor (CAR) T Cell Therapy, in Adult Patients with Relapsed/ Refractory Acute Lymphoblastic Leukemia (R/R ALL): Outcomes in Patients Who Were Treated with Prior Blinatumomab in ZUMA-3 [Abstract ALL-128]. Clinical lymphoma, myeloma & leukemia 2018;18 (Supplement 1):S184.
- [Result] Shah BD, Oluwole OO, Baer MR, Bishop MR, Holmes H, Schiller GJ, et al. Outcomes of Patients Treated With Prior Blinatumomab in ZUMA-3, a Study of KTE-C19, an Anti-CD19 Chimeric Antigen Receptor T Cell Therapy, in Adult Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia. ASCO; 2018 01-05 June; Chicago, IL.
- [Result] Shah BD, Stock W, Wierda WG, Oluwole O, Holmes H, Schiller GJ, et al. Phase 1 Results of ZUMA-3: KTE-C19, an Anti-CD19 Chimeric Antigen Receptor (CAR) T Cell Therapy, in Adult Patients with Relapsed/Refractory Acute Lymphoblastic Leukemia (R/R ALL) [Abstract 612]. Blood 2017;130 (Supplement 1):888.
- [Result] Shah BD, Wierda WG, Schiller GJ, Bishop MR, Castro JE, Sabatino M, et al. Updated results from ZUMA- 3, a phase 1/2 study of KTE-C19 chimeric antigen receptor (CAR) T cell therapy, in adults with high-burden relapsed/refractory acute lymphoblastic leukemia (R/R ALL) [Abstract 3024]. American Society of Clinical Oncology (ASCO) Annual Meeting; 2017 02-06 June; Chicago, Illinois.
- [Result] Wierda WG, Bishop MR, Oluwole O, Logan AC, Baer MR, Donnellan WB, et al. Updated Phase 1 Results of Zuma-3: Kte-X19, an Anti-CD19 Chimeric Antigen Receptor T Cell Therapy, in Adult Patients with Relapsed/Refractory Acute Lymphoblastic Leukemia [Abstract 256]. Biol Blood Marrow Transplant 2019;25 (3):S185.
- [Result] Wierda WG, Bishop MR, Oluwole OO, Logan AC, Baer MR, Donnellan WB, et al. Updated Phase 1 Results of Zuma-3: Kte-C19, an Anti-CD19 Chimeric Antigen Receptor T Cell Therapy, in Adult Patients with Relapsed/Refractory Acute Lymphoblastic Leukemia [Abstract]. Blood 2018;132 (Supplement 1):897.
- [Result] Shah BD, Bishop MR, Oluwole OO, Logan AC, Baer MR, Donnellan WB, O'Dwyer KM, Holmes H, Arellano ML, Ghobadi A, Pagel JM, Lin Y, Cassaday RD, Park JH, Abedi M, Castro JE, DeAngelo DJ, Malone AK, Mawad R, Schiller GJ, Rossi JM, Bot A, Shen T, Goyal L, Jain RK, Vezan R, Wierda WG. KTE-X19 anti-CD19 CAR T-cell therapy in adult relapsed/refractory acute lymphoblastic leukemia: ZUMA-3 phase 1 results. Blood. 2021 Jul 8;138(1):11-22. doi: 10.1182/blood.2020009098. PMID 33827116
- [Result] Shah BD, Ghobadi A, Oluwole OO, Logan AC, Boissel N, Cassaday RD, Leguay T, Bishop MR, Topp MS, Tzachanis D, O'Dwyer KM, Arellano ML, Lin Y, Baer MR, Schiller GJ, Park JH, Subklewe M, Abedi M, Minnema MC, Wierda WG, DeAngelo DJ, Stiff P, Jeyakumar D, Feng C, Dong J, Shen T, Milletti F, Rossi JM, Vezan R, Masouleh BK, Houot R. KTE-X19 for relapsed or refractory adult B-cell acute lymphoblastic leukaemia: phase 2 results of the single-arm, open-label, multicentre ZUMA-3 study. Lancet. 2021 Aug 7;398(10299):491-502. doi: 10.1016/S0140-6736(21)01222-8. Epub 2021 Jun 4. PMID 34097852
- [Derived] Shah BD, Ghobadi A, Oluwole OO, Logan AC, Boissel N, Cassaday RD, Leguay T, Bishop MR, Topp MS, Tzachanis D, O'Dwyer KM, Arellano ML, Lin Y, Baer MR, Schiller GJ, Park JH, Subklewe M, Abedi M, Minnema MC, Wierda WG, DeAngelo DJ, Stiff P, Jeyakumar D, Dong J, Adhikary S, Zhou L, Schuberth PC, Faghmous I, Masouleh BK, Houot R. Two-year follow-up of KTE-X19 in patients with relapsed or refractory adult B-cell acute lymphoblastic leukemia in ZUMA-3 and its contextualization with SCHOLAR-3, an external historical control study. J Hematol Oncol. 2022 Dec 10;15(1):170. doi: 10.1186/s13045-022-01379-0. PMID 36494725
- [Derived] Shah BD, Smith NJ, Feng C, Jeyakumar S, Castaigne JG, Faghmous I, Masouleh BK, Malone DC, Bishop MR. Cost-Effectiveness of KTE-X19 for Adults with Relapsed/Refractory B-Cell Acute Lymphoblastic Leukemia in the United States. Adv Ther. 2022 Aug;39(8):3678-3695. doi: 10.1007/s12325-022-02201-6. Epub 2022 Jun 21. PMID 35727476
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KTE-C19-103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in France, Germany, the Netherlands, and the United States.
Pre-assignment Details: 173 participants were screened. Bridging therapy was recommended for all participants particularly those participants with high disease burden at baseline (M3 marrow [> 25% leukemic blasts] or ≥ 1,000 blasts/mm^3 in the peripheral circulation) to control participant's disease post apheresis/enrollment and prior to conditioning chemotherapy.
Groups:
- Phase 1: 2 x 10^6 Anti-CD19 CAR T Cells/kg: Participants with relapsed or refractory B-precursor acute lymphoblastic leukemia (r/r B-ALL) received conditioning chemotherapy (fludarabine 25 mg/m^2 intravenously [IV] over 30 minutes on Day -4, Day -3, and Day -2 and cyclophosphamide 900 mg/m^2 IV over 60 minutes on Day -2) followed by a single infusion of brexucabtagene autoleucel (KTE-X19) chimeric antigen receptor (CAR) transduced autologous T cells administered IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of body weight on Day 0. For participants weighing > 100 kg, a maximum flat dose of 2 x 10^8 anti-CD19 CAR T cells/kg of body weight was administered.
- Phase 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg; Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg: Participants with r/r B-ALL received conditioning chemotherapy (fludarabine 25 mg/m^2 IV over 30 minutes on Day -4, Day -3, and Day -2 and cyclophosphamide 900 mg/m^2 IV over 60 minutes on Day -2) followed by a single infusion of brexucabtagene autoleucel CAR transduced autologous T cells administered IV at a target dose of 1 x 10^6 anti-CD19 CAR T cells/kg of body weight on Day 0. For participants weighing > 100 kg, a maximum flat dose of 1 x 10^8 anti-CD19 CAR T cells/kg of body weight was administered.
- Phase 1: 0.5 x 10^6 Anti-CD19 CAR T Cells/kg: Participants with r/r B-ALL received conditioning chemotherapy (fludarabine 25 mg/m^2 IV over 30 minutes on Day -4, Day -3, and Day -2 and cyclophosphamide 900 mg/m^2 IV over 60 minutes on Day -2) followed by a single infusion of brexucabtagene autoleucel CAR transduced autologous T cells administered IV at a target dose of 0.5 x 10^6 anti-CD19 CAR T cells/kg of body weight on Day 0. For participants weighing > 100 kg, a maximum flat dose of 0.5 x 10^8 anti-CD19 CAR T cells/kg of body weight was administered.
Period: Overall Study
Arm/Group | Phase 1: 2 x 10^6 Anti-CD19 CAR T Cells/kg | Phase 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Phase 1: 0.5 x 10^6 Anti-CD19 CAR T Cells/kg | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Started | 6 | 28 | 20 | 71
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 28 | 20 | 71
Not completed — Death | 6 | 14 | 11 | 29
Not completed — Full consent withdrawn | 0 | 1 | 0 | 8
Not completed — Lost to Follow-up | 0 | 2 | 2 | 2
Not completed — Enrolled but did not Initiate KTE-X19 | 0 | 5 | 4 | 16
Not completed — Rolled over or consented to a long term follow-up (LFTU) study | 0 | 4 | 2 | 15
Not completed — Reason not specified | 0 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants treated with any dose of brexucabtagene autoleucel.
Groups:
- Phase 1: 2 x 10^6 Anti-CD19 CAR T Cells/kg: Participants with r/r B-ALL received conditioning chemotherapy (fludarabine 25 mg/m^2 IV over 30 minutes on Day -4, Day -3, and Day -2 and cyclophosphamide 900 mg/m^2 IV over 60 minutes on Day -2) followed by a single infusion of brexucabtagene autoleucel CAR transduced autologous T cells administered IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of body weight on Day 0. For participants weighing > 100 kg, a maximum flat dose of 2 x 10^8 anti-CD19 CAR T cells/kg of body weight was administered.
- Total: Total of all reporting groups
Arm/Group | Phase 1: 2 x 10^6 Anti-CD19 CAR T Cells/kg | Phase 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Phase 1: 0.5 x 10^6 Anti-CD19 CAR T Cells/kg | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Total
Number analyzed (Participants) | 6 | 23 | 16 | 55 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (13.8) | 46 (17.6) | 46 (16.7) | 42 (16.1) | 43 (16.3)
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 1
  Between 18 and 65 years | 6 | 18 | 13 | 47 | 84
  >=65 years | 0 | 4 | 3 | 8 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 14 | 8 | 22 | 45
  Male | 5 | 9 | 8 | 33 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 3 | 11 | 3 | 11 | 28
  Ethnicity: Not Hispanic or Latino | 3 | 12 | 13 | 42 | 70
  Ethnicity: Not collected | 0 | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Race: Asian | 1 | 2 | 0 | 3 | 6
  Race: Black or African American | 0 | 0 | 0 | 1 | 1
  Race: White | 4 | 19 | 16 | 37 | 76
  Race: Other or More Than One Race | 1 | 1 | 0 | 9 | 11
  Race: Not collected | 0 | 0 | 0 | 4 | 4
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  France | 0 | 0 | 0 | 10 | 10
  Germany | 0 | 0 | 0 | 3 | 3
  Netherlands | 0 | 0 | 0 | 1 | 1
  United States | 6 | 23 | 16 | 41 | 86

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs)
Description: DLT is drug-related events with onset within first 28 days following infusion:
  * Grade (GR) 4 hematologic toxicity lasting more than 30 days (except lymphopenia) if not attributable to underlying disease
  * All drug-related GR 3 lasting for > 7 days or 4 non-hematologic toxicities regardless of duration (except: aphasia/dysphasia or confusion/cognitive disturbance which resolves to at least GR 1/baseline within 2 weeks or baseline within 4 weeks, fever GR 3/ 4, immediate hypersensitivity reactions within 2 hours of drug infusion that are reversible ≤ GR 2 within 24 hours, renal toxicity which requires dialysis for ≤ 7 days, intubation for airway protection if ≤ 7 days, tumor lysis syndrome, GR 3 liver function test elevation, provided there is resolution to ≤ GR 2 within 14 days, GR 4 transient serum hepatic enzyme abnormalities provided there is resolution to ≤ GR 3 within < 72 hours, hypogammaglobulinemia GR 3/ 4 and GR 3 nausea and/or anorexia).
Time Frame: First infusion date of brexucabtagene autoleucel up to 28 days. Participants were evaluated in specified period but GR4 hematologic toxicity (specified in description) having onset in this period were further observed for 30 days for confirmation
Population: DLT-Evaluable Analysis Set included first 3 participants in Phase 1 treated with target brexucabtagene autoleucel dose and followed for at least 28 days. Only participants from Phase 1: 2 X 10^6 Anti-CD19 CAR T Cells/kg were pre-specified to be assessed for this Outcome Measure.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: 2 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 3
percentage of participants | 0

2. Primary Outcome: Phase 2: Overall Complete Remission (OCR) Rate (Complete Remission [CR]+ Complete Remission With Incomplete Hematologic Recovery [CRi]) as Assessed Per Independent Review
Description: OCR rate:percentage of participants achieving CR+CRi.CR: ≤5% blasts by morphology in bone marrow(BM);absolute neutrophil count(ANC)≥1000/microliters (μL) and platelets(Plt) ≥100000/μL in peripheral blood(PB);central nervous system extramedullary disease(CNS EMD) of CNS-1(no detectable leukemia in cerebrospinal fluid[CSF]);Non-CNS baselineEMD:if present(images shows CR),if no(images not needed),if performed shows negative positron emission tomography(PET) baseline,baseline lesions shows CR as disappearance of measurable and nonmeasurable nodal lesions(Nodal masses >1.5 cm in greatest transverse diameter[GTD] at baseline have regressed to ≤l.5 cm GTD,nodes that were 1.1 to 1.5 cm[long axis] and >1.0 cm[short axis] have decreased to 1.0 cm in their short axis, spleen and/or liver must be normal size) and no new lesions.CRi:all CR criteria except in PB ANC≥1000/μL and Plt<100000/μL or ANC<1000/μL and Plt ≥100000/μL.95% confidence interval (CI) was calculated by Clopper-Pearson method.
Time Frame: First infusion date of brexucabtagene autoleucel (Phase 2) up to 3.7 years
Population: The modified Intent-to-Treat (mITT) Analysis Set included all enrolled participants treated with brexucabtagene autoleucel in Phase 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
percentage of participants | 70.9 [57 to 82]

3. Secondary Outcome: Phase 2: Minimum Residual Disease (MRD) Negative Remission Rate
Description: MRD was assessed utilizing multicolor flow cytometry to detect residual cancerous cells with a sensitivity of 10^-4. MRD negative remission was defined as MRD < 10^-4 threshold. Percentage of participants with MRD negative remission was reported. 95% CI was calculated by Clopper-Pearson method.
Time Frame: First infusion date of brexucabtagene autoleucel (Phase 2) up to 3.7 years
Population: Participants in mITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
percentage of participants | 76 [63 to 87]

4. Secondary Outcome: Phase 2: Complete Remission (CR) Rate Per Independent Review
Description: CR: ≤ 5% blasts by morphology in BM; ANC ≥ 1000/µL and Plt ≥ 100000/µL in PB; CNS EMD of CNS-1 (no detectable leukemia in CSF); Non-CNS EMD: if baseline EMD present (images must show CR), if no baseline EMD (then images not required), but if performed should show negative PET baseline, baseline lesions must show CR as disappearance of measurable and nonmeasurable nodal lesions (Nodal masses > 1.5 cm in GTD at baseline must have regressed to ≤ l.5 cm GTD, nodes that were 1.1 to 1.5 cm [long axis] and > 1.0 cm [short axis] must have decreased to 1.0 cm in their short axis, spleen and/or liver must be normal size) and no new lesions. Percentage of participants with CR was reported. 95% CI was calculated by Clopper-Pearson method.
Time Frame: First infusion date of brexucabtagene autoleucel (Phase 2) up to 3.7 years
Population: Participants in mITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
percentage of participants | 56.4 [42 to 70]

5. Secondary Outcome: Phase 2: Complete Remission With Incomplete Hematologic Recovery (CRi) Rate Per Independent Review
Description: CRi: ≤ 5% blasts by morphology in BM; ANC ≥ 1000/µL and Plt < 100000/µL or ANC < 1000/µL and Plt ≥ 100000/µL in PB; CNS EMD of CNS-1 (no detectable leukemia in CSF); Non-CNS EMD: if baseline EMD present (images must show CR), if no baseline EMD (then images not required), but if performed should show negative PET baseline, baseline lesions must show CR as disappearance of measurable and nonmeasurable nodal lesions (Nodal masses > 1.5 cm in GTD at baseline must have regressed to ≤ l.5 cm GTD, nodes that were 1.1 to 1.5 cm [long axis] and > 1.0 cm [short axis] must have decreased to 1.0 cm in their short axis, spleen and/or liver must be normal size, if tested) and no new lesions. Percentage of participants with CRi was reported. 95% CI was calculated by Clopper-Pearson method.
Time Frame: First infusion date of brexucabtagene autoleucel (Phase 2) up to 3.7 years
Population: Participants in mITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
percentage of participants | 14.5 [6 to 27]

6. Secondary Outcome: Phase 2: Duration of Remission (DOR) Per Independent Review
Description: DOR was defined as the time from first CR or CRi to relapse or any death in the absence of documented relapse. CR and CRi are defined in Outcome Measures 4 and 5. Relapse: ≤ 5% blasts by morphology in BM; or circulating leukemia present in PB; or CNS EMD of CNS-2 (detectable CSF blast cells in a sample of CSF with < 5 white blood cells [WBCs] per mm^3 with neurological changes) or CNS-3 (detectable CSF blast cells in a sample of CSF with ≥ 5 WBCs per mm^3 with or without neurological changes); or progressive disease (PD): at least one of the following (≥ 50% increase from nadir in the sum of the products of at least two lymph nodes, or if a single node is involved at least a 50% increase in the product of the diameters of this one node; at least a 50% increase in the longest diameter of any single previously identified node more than 1 cm in its short axis; ≥ 50% increase in size of splenic, hepatic or any other non-nodal lesion). Kaplan-Meier (KM) estimates was used for analyses.
Time Frame: From first CR or CRi (Phase 2) up to 3.7 years
Population: Participants in mITT Analysis Set with overall complete remission (CR or CRi ) were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 39
months | 14.6 [9.4 to 24.1]

7. Secondary Outcome: Phase 2: OCR Rate (CR + CRi) Per Investigator Review
Description: OCR rate: percentage of participants achieving CR+CRi. CR: ≤ 5% blasts by morphology in BM; ANC ≥1000/µL and Plt ≥ 100000/µL in PB; CNS EMD of CNS-1 (no detectable leukemia in CSF); Non-CNS EMD: if baseline EMD present (images must show CR), if no baseline EMD (then images not required), but if performed should show negative PET baseline, baseline lesions must show CR as disappearance of measurable and nonmeasurable nodal lesions (Nodal masses >1.5 cm in GTD at baseline must have regressed to ≤l.5 cm GTD, nodes that were 1.1 to 1.5 cm [long axis] and >1.0 cm [short axis] must have decreased to 1.0 cm in their short axis, spleen and/or liver must be normal size, if tested) and no new lesions. CRi: all CR criteria except in PB ANC ≥1000/µL and Plt <100000/µL or ANC <1000/µL and Plt ≥100000/µL. 95% CI was calculated by Clopper-Pearson method.
Time Frame: First infusion date of brexucabtagene autoleucel (Phase 2) up to 5 years
Population: Participants in mITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
percentage of participants | 72.7 [59 to 84]

8. Secondary Outcome: Phase 2: Percentage of Participants With Allogeneic Stem Cell Transplant (Allo-SCT)
Time Frame: First infusion date of brexucabtagene autoleucel (Phase 2) up to 5 years
Population: Participants in mITT Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
percentage of participants | 20

9. Secondary Outcome: Phase 2: MRD Negative Remission Rate Among Complete Remission (CR) Participants
Description: Percentage of participants with MRD negative remission among CR participants was reported. MRD was assessed utilizing multicolor flow cytometry to detect residual cancerous cells with a sensitivity of 10^-4. MRD negative remission was defined as MRD < 10^-4 threshold. CR: ≤5% blasts by morphology in BM; ANC ≥ 1000/µL and Plt ≥ 100000/µL in PB; CNS EMD of CNS-1 (no detectable leukemia in CSF); Non-CNS EMD: if baseline EMD present (images must show CR), if no baseline EMD (then images not required), but if performed should show negative PET baseline, baseline lesions must show CR as disappearance of measurable and nonmeasurable nodal lesions (Nodal masses > 1.5 cm in GTD at baseline must have regressed to ≤ l.5 cm GTD, nodes that were 1.1 to 1.5 cm [long axis] and > 1.0 cm [short axis] must have decreased to 1.0 cm in their short axis, spleen and/or liver must be normal size) and no new lesions. 95% CI was calculated by Clopper-Pearson method.
Time Frame: First infusion date of brexucabtagene autoleucel (Phase 2) up to 3.7 years
Population: Participants in mITT Analysis Set with CR were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 31
percentage of participants | 97 [83 to 100]

10. Secondary Outcome: Phase 2: MRD Negative Remission Rate Among Complete Remission With Incomplete Hematologic Recovery (CRi) Participants
Description: Percentage of participants with MRD negative remission among CRi participants was reported. MRD was assessed utilizing multicolor flow cytometry to detect residual cancerous cells with a sensitivity of 10^-4. MRD negative remission was defined as MRD < 10^-4 threshold. CRi: ≤ 5% blasts by morphology in BM; ANC ≥ 1000/µL and Plt < 100000/µL or ANC < 1000/µL and Plt ≥ 100000/µL in PB; CNS EMD of CNS-1 (no detectable leukemia in CSF); Non-CNS EMD: if baseline EMD present (images must show CR), if no baseline EMD (then images not required), but if performed should show negative PET baseline, baseline lesions must show CR as disappearance of measurable and nonmeasurable nodal lesions (Nodal masses >1.5 cm in GTD at baseline must have regressed to ≤l.5 cm GTD, nodes that were 1.1 to 1.5 cm [long axis] and >1.0 cm [short axis] must have decreased to 1.0 cm in their short axis, spleen and/or liver must be normal size) and no new lesions. 95% CI was calculated by Clopper-Pearson method.
Time Frame: First infusion date of brexucabtagene autoleucel (Phase 2) up to 3.7 years
Population: Participants in mITT Analysis Set with CRi were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 8
percentage of participants | 100 [63 to 100]

11. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time from brexucabtagene autoleucel infusion to the date of death from any cause. Participants who had not died by the analysis data cutoff date were censored at their last contact date. KM estimates was used for analyses.
Time Frame: First infusion date of brexucabtagene autoleucel (Phase 2) up to 5 years
Population: Participants in mITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
months | 26.0 [16.2 to NA] — Upper limit of confidence interval was not estimable due to insufficient number of events.

12. Secondary Outcome: Phase 2: Relapse-free Survival (RFS)
Description: RFS: time from brexucabtagene autoleucel infusion to date of disease relapse or death from any cause. Participants not meeting criteria for relapse by the analysis data cutoff date were censored at their last evaluable disease assessment date. Participants who had not achieved a CR or CRi at analysis data cutoff were evaluated as an RFS event at Day 0. CR and CRi are defined in Outcome Measures 4 and 5. Relapse is defined in Outcome Measure 6. KM estimates was used for analyses.
Time Frame: First infusion date of brexucabtagene autoleucel (Phase 2) up to 3.7 years
Population: Participants in mITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
months | 11.6 [2.7 to 20.5]

13. Secondary Outcome: Phase 2: Percentage of Participants Experiencing Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant after brexucabtagene autoleucel infusion, which did not necessarily have a causal relationship with the treatment. An AE could therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. TEAEs included all AEs with onset on or after initiation of the brexucabtagene autoleucel infusion.
Time Frame: Up to 5 years
Population: The Safety Analysis Set included all participants treated with any dose of brexucabtagene autoleucel.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
percentage of participants | 100

14. Secondary Outcome: Phase 2: Number of Participants Experiencing Laboratory Toxicity Grade 3 or Higher TEAEs Resulting From Increased Parameter Value
Description: Grading categories are determined by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Grade 1: mild, Grade 2: moderate, Grade 3: severe or medically significant, Grade 4: life-threatening.
Time Frame: Up to 5 years
Population: Participants in Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
Participants
  Hematology: Lymphocytes | 1
  Hematology: Leukocytes | 4
  Hematology: Hemoglobin | 0
  Hematology: Neutrophils | 0
  Hematology: Platelets | 0
  Chemistry: Creatinine | 4
  Chemistry: Glucose | 13
  Chemistry: Aspartate Aminotransferase | 14
  Chemistry: Alanine Aminotransferase | 17
  Chemistry: Bilirubin | 5
  Chemistry: Alkaline Phosphatase | 3
  Chemistry: Direct Bilirubin | 8
  Chemistry: Urate | 12
  Chemistry: Sodium | 1
  Chemistry: Potassium | 2
  Chemistry: Magnesium | 3
  Chemistry: Calcium | 0
  Chemistry: Albumin | 0
  Chemistry: Phosphate | 0

15. Secondary Outcome: Phase 2: Number of Participants Experiencing Laboratory Toxicity Grade 3 or Higher TEAEs Resulting From Decreased Parameter Value
Description: Grading categories are determined by CTCAE version 4.03. Grade 1: mild, Grade 2: moderate, Grade 3: severe or medically significant, Grade 4: life-threatening.
Time Frame: Up to 5 years
Population: Participants in Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
Participants
  Hematology: Hemoglobin | 42
  Hematology: Leukocytes | 54
  Hematology: Platelets | 46
  Hematology: Lymphocytes | 52
  Hematology: Neutrophils | 53
  Chemistry: Calcium | 9
  Chemistry: Albumin | 5
  Chemistry: Phosphate | 27
  Chemistry: Magnesium | 0
  Chemistry: Sodium | 11
  Chemistry: Potassium | 7
  Chemistry: Glucose | 0
  Chemistry: Alanine Aminotransferase | 0
  Chemistry: Alkaline Phosphatase | 0
  Chemistry: Aspartate Aminotransferase | 0
  Chemistry: Bilirubin | 0
  Chemistry: Creatinine | 0
  Chemistry: Direct Bilirubin | 0
  Chemistry: Urate | 0

16. Secondary Outcome: Phase 2: Percentage of Participants With Anti-KTE-X19 Antibodies
Time Frame: First infusion date of brexucabtagene autoleucel (Phase 2) up to 2.7 years
Population: Participants in Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 55
percentage of participants | 7

17. Secondary Outcome: Phase 2: Number of Participants With 5-Level European Quality of Life-5 Dimensions (EQ-5D-5L): Health Utility Index Scale
Description: The EQ-5D-5 levels(EQ-5D-5L)is a standardized measure of health status of the participant that provides a simple, generic measure of health for clinical and economic appraisal.It is a self-reported questionnaire used to assess the overall health status of participant scoring 5 dimensions of health: mobility,self-care,usual activities,pain/discomfort and anxiety/depression.Each dimension has 5 levels:no problems,slight problems,moderate problems,severe problems,and extreme problems.EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by a formula that attaches values (called QOL utilities)to each of the levels in each dimension.EQ-5D Summary Index values range from -0.11(worst health) to 1.00(perfect health).This decision results in a 1-digit number that shows the level for that dimension. The digits for 5 dimensions can be combined to 5-digit number that show the participant's health.Higher scores of EQ-5D-5L indicate better health.
Time Frame: Baseline, Day 28, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, and Month 24
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 51
Participants
  Baseline: Mobility (No problem) | 39
  Baseline: Mobility (Slight problem) | 7
  Baseline: Mobility (Moderate problem) | 4
  Baseline: Mobility (Severe problem) | 1
  Baseline: Mobility (Unable to walk) | 0
  Day 28: Mobility (No problem): number analyzed (Participants) | 42
  Day 28: Mobility (No problem) | 19
  Day 28: Mobility (Slight problem): number analyzed (Participants) | 42
  Day 28: Mobility (Slight problem) | 10
  Day 28: Mobility (Moderate problem): number analyzed (Participants) | 42
  Day 28: Mobility (Moderate problem) | 9
  Day 28: Mobility (Severe problem): number analyzed (Participants) | 42
  Day 28: Mobility (Severe problem) | 1
  Day 28: Mobility (Unable to walk): number analyzed (Participants) | 42
  Day 28: Mobility (Unable to walk) | 3
  Month 3: Mobility (No problem): number analyzed (Participants) | 26
  Month 3: Mobility (No problem) | 19
  Month 3: Mobility (Slight problem): number analyzed (Participants) | 26
  Month 3: Mobility (Slight problem) | 5
  Month 3: Mobility (Moderate problem): number analyzed (Participants) | 26
  Month 3: Mobility (Moderate problem) | 1
  Month 3: Mobility (Severe problem): number analyzed (Participants) | 26
  Month 3: Mobility (Severe problem) | 0
  Month 3: Mobility (Unable to walk): number analyzed (Participants) | 26
  Month 3: Mobility (Unable to walk) | 1
  Month 6: Mobility (No problem): number analyzed (Participants) | 25
  Month 6: Mobility (No problem) | 16
  Month 6: Mobility (Slight problem): number analyzed (Participants) | 25
  Month 6: Mobility (Slight problem) | 6
  Month 6: Mobility (Moderate problem): number analyzed (Participants) | 25
  Month 6: Mobility (Moderate problem) | 2
  Month 6: Mobility (Severe problem): number analyzed (Participants) | 25
  Month 6: Mobility (Severe problem) | 0
  Month 6: Mobility (Unable to walk): number analyzed (Participants) | 25
  Month 6: Mobility (Unable to walk) | 1
  Month 9: Mobility (No problem): number analyzed (Participants) | 10
  Month 9: Mobility (No problem) | 8
  Month 9: Mobility (Slight problem): number analyzed (Participants) | 10
  Month 9: Mobility (Slight problem) | 1
  Month 9: Mobility (Moderate problem): number analyzed (Participants) | 10
  Month 9: Mobility (Moderate problem) | 0
  Month 9: Mobility (Severe problem): number analyzed (Participants) | 10
  Month 9: Mobility (Severe problem) | 0
  Month 9: Mobility (Unable to walk): number analyzed (Participants) | 10
  Month 9: Mobility (Unable to walk) | 1
  Month 12: Mobility (No problem): number analyzed (Participants) | 14
  Month 12: Mobility (No problem) | 11
  Month 12: Mobility (Slight problem): number analyzed (Participants) | 14
  Month 12: Mobility (Slight problem) | 3
  Month 12: Mobility (Moderate problem): number analyzed (Participants) | 14
  Month 12: Mobility (Moderate problem) | 0
  Month 12: Mobility (Severe problem): number analyzed (Participants) | 14
  Month 12: Mobility (Severe problem) | 0
  Month 12: Mobility (Unable to walk): number analyzed (Participants) | 14
  Month 12: Mobility (Unable to walk) | 0
  Month 15: Mobility (No problem): number analyzed (Participants) | 10
  Month 15: Mobility (No problem) | 7
  Month 15: Mobility (Slight problem): number analyzed (Participants) | 10
  Month 15: Mobility (Slight problem) | 2
  Month 15: Mobility (Moderate problem): number analyzed (Participants) | 10
  Month 15: Mobility (Moderate problem) | 1
  Month 15: Mobility (Severity problem): number analyzed (Participants) | 10
  Month 15: Mobility (Severity problem) | 0
  Month 15: Mobility (Unable to walk): number analyzed (Participants) | 10
  Month 15: Mobility (Unable to walk) | 0
  Month 18: Mobility (No problem): number analyzed (Participants) | 4
  Month 18: Mobility (No problem) | 3
  Month 18: Mobility (Slight problem): number analyzed (Participants) | 4
  Month 18: Mobility (Slight problem) | 1
  Month 18: Mobility (Moderate problem): number analyzed (Participants) | 4
  Month 18: Mobility (Moderate problem) | 0
  Month 18: Mobility (Severe problem): number analyzed (Participants) | 4
  Month 18: Mobility (Severe problem) | 0
  Month 18: Mobility (Unable to walk): number analyzed (Participants) | 4
  Month 18: Mobility (Unable to walk) | 0
  Month 24: Mobility (No problem): number analyzed (Participants) | 4
  Month 24: Mobility (No problem) | 3
  Month 24: Mobility (Slight problem): number analyzed (Participants) | 4
  Month 24: Mobility (Slight problem) | 1
  Month 24: Mobility (Moderate problem): number analyzed (Participants) | 4
  Month 24: Mobility (Moderate problem) | 0
  Month 24: Mobility (Severe problem): number analyzed (Participants) | 4
  Month 24: Mobility (Severe problem) | 0
  Month 24: Mobility (Unable to Walk): number analyzed (Participants) | 4
  Month 24: Mobility (Unable to Walk) | 0
  Baseline: Self-care (No problem) | 44
  Baseline: Self-care (Slight problem) | 5
  Baseline: Self-care (Moderate problem) | 1
  Baseline: Self-care (Severe problem) | 1
  Baseline: Self-care (Unable to wash or dress) | 0
  Day 28: Self-care (No problem): number analyzed (Participants) | 42
  Day 28: Self-care (No problem) | 31
  Day 28: Self-care (Slight problem): number analyzed (Participants) | 42
  Day 28: Self-care (Slight problem) | 6
  Day 28: Self-care (Moderate problem): number analyzed (Participants) | 42
  Day 28: Self-care (Moderate problem) | 1
  Day 28: Self-care (Severe problem): number analyzed (Participants) | 42
  Day 28: Self-care (Severe problem) | 2
  Day 28: Self-care (Unable to wash or dress): number analyzed (Participants) | 42
  Day 28: Self-care (Unable to wash or dress) | 2
  Month 3: Self-care (No problem): number analyzed (Participants) | 25
  Month 3: Self-care (No problem) | 23
  Month 3: Self-care (Slight problem): number analyzed (Participants) | 25
  Month 3: Self-care (Slight problem) | 1
  Month 3: Self-care (Moderate problem): number analyzed (Participants) | 25
  Month 3: Self-care (Moderate problem) | 1
  Month 3: Self-care (Severe problem): number analyzed (Participants) | 25
  Month 3: Self-care (Severe problem) | 0
  Month 3: Self-care (Unable to wash or dress): number analyzed (Participants) | 25
  Month 3: Self-care (Unable to wash or dress) | 0
  Month 6: Self-care (No problem): number analyzed (Participants) | 25
  Month 6: Self-care (No problem) | 23
  Month 6: Self-care (Slight problem) | 0
  Month 6: Self-care (Moderate problem) | 1
  Month 6: Self-care (Severe problem) | 1
  Month 6: Self-care (Unable to wash or dress): number analyzed (Participants) | 10
  Month 6: Self-care (Unable to wash or dress) | 0
  Month 9: Self-care (No problem): number analyzed (Participants) | 10
  Month 9: Self-care (No problem) | 9
  Month 9: Self-care (Slight problem): number analyzed (Participants) | 10
  Month 9: Self-care (Slight problem) | 0
  Month 9: Self-care (Moderate problem): number analyzed (Participants) | 10
  Month 9: Self-care (Moderate problem) | 0
  Month 9: Self-care (Severe problem): number analyzed (Participants) | 10
  Month 9: Self-care (Severe problem) | 1
  Month 9: Self-care (Unable to wash or dress) | 0
  Month 12: Self-care (No problem): number analyzed (Participants) | 14
  Month 12: Self-care (No problem) | 14
  Month 12: Self-care (Slight problem): number analyzed (Participants) | 14
  Month 12: Self-care (Slight problem) | 0
  Month 12: Self-care (Moderate problem): number analyzed (Participants) | 14
  Month 12: Self-care (Moderate problem) | 0
  Month 12: Self-care (Severe problem): number analyzed (Participants) | 14
  Month 12: Self-care (Severe problem) | 0
  Month 12: Self-care (Unable to wash or dress): number analyzed (Participants) | 14
  Month 12: Self-care (Unable to wash or dress) | 0
  Month 15: Self-care (No problem): number analyzed (Participants) | 10
  Month 15: Self-care (No problem) | 10
  Month 15: Self-care (Slight problem): number analyzed (Participants) | 10
  Month 15: Self-care (Slight problem) | 0
  Month 15: Self-care (Moderate problem): number analyzed (Participants) | 10
  Month 15: Self-care (Moderate problem) | 0
  Month 15: Self-care (Severe problem): number analyzed (Participants) | 10
  Month 15: Self-care (Severe problem) | 0
  Month 15: Self-care (Unable to wash or dress): number analyzed (Participants) | 10
  Month 15: Self-care (Unable to wash or dress) | 0
  Month 18: Self-care (No problem): number analyzed (Participants) | 4
  Month 18: Self-care (No problem) | 4
  Month 18: Self-care (Slight problem): number analyzed (Participants) | 4
  Month 18: Self-care (Slight problem) | 0
  Month 18: Self-care (Moderate problem): number analyzed (Participants) | 4
  Month 18: Self-care (Moderate problem) | 0
  Month 18: Self-care (Severe problem): number analyzed (Participants) | 4
  Month 18: Self-care (Severe problem) | 0
  Month 18: Self-care (Unable to wash or dress): number analyzed (Participants) | 4
  Month 18: Self-care (Unable to wash or dress) | 0
  Month 24: Self-care (No problem): number analyzed (Participants) | 4
  Month 24: Self-care (No problem) | 4
  Month 24: Self-care (Slight problem): number analyzed (Participants) | 4
  Month 24: Self-care (Slight problem) | 0
  Month 24: Self-care (Moderate problem): number analyzed (Participants) | 4
  Month 24: Self-care (Moderate problem) | 0
  Month 24: Self-care (Severe problem): number analyzed (Participants) | 4
  Month 24: Self-care (Severe problem) | 0
  Month 24: Self-care (Unable to wash or dress): number analyzed (Participants) | 4
  Month 24: Self-care (Unable to wash or dress) | 0
  Baseline: Usual activities (No problem) | 24
  Baseline: Usual activities (Slight problem) | 14
  Baseline: Usual activities (Moderate problem) | 9
  Baseline: Usual activities (Severe problem) | 3
  Baseline: Usual activities (Unable to do usual activities) | 1
  Day 28: Usual activities (No problem): number analyzed (Participants) | 42
  Day 28: Usual activities (No problem) | 17
  Day 28: Usual activities (Slight problem): number analyzed (Participants) | 42
  Day 28: Usual activities (Slight problem) | 13
  Day 28: Usual activities (Moderate problem): number analyzed (Participants) | 42
  Day 28: Usual activities (Moderate problem) | 8
  Day 28: Usual activities (Severe problem): number analyzed (Participants) | 42
  Day 28: Usual activities (Severe problem) | 3
  Day 28: Usual activities (Unable to do usual activities): number analyzed (Participants) | 42
  Day 28: Usual activities (Unable to do usual activities) | 1
  Month 3: Usual activities (No problem): number analyzed (Participants) | 25
  Month 3: Usual activities (No problem) | 14
  Month 3: Usual activities (Slight problem): number analyzed (Participants) | 25
  Month 3: Usual activities (Slight problem) | 9
  Month 3: Usual activities (Moderate problem): number analyzed (Participants) | 25
  Month 3: Usual activities (Moderate problem) | 1
  Month 3: Usual activities (Severe problem): number analyzed (Participants) | 25
  Month 3: Usual activities (Severe problem) | 1
  Month 3: Usual activities (Unable to do usual activities): number analyzed (Participants) | 25
  Month 3: Usual activities (Unable to do usual activities) | 0
  Month 6: Usual activities (No problem): number analyzed (Participants) | 25
  Month 6: Usual activities (No problem) | 17
  Month 6: Usual activities (Slight problem): number analyzed (Participants) | 25
  Month 6: Usual activities (Slight problem) | 4
  Month 6: Usual activities (Moderate problem): number analyzed (Participants) | 25
  Month 6: Usual activities (Moderate problem) | 2
  Month 6: Usual activities (Severe problem): number analyzed (Participants) | 25
  Month 6: Usual activities (Severe problem) | 2
  Month 6: Usual activities (Unable to do usual activities): number analyzed (Participants) | 25
  Month 6: Usual activities (Unable to do usual activities) | 0
  Month 9: Usual activities (No problem): number analyzed (Participants) | 10
  Month 9: Usual activities (No problem) | 9
  Month 9: Usual activities (Slight problem): number analyzed (Participants) | 10
  Month 9: Usual activities (Slight problem) | 0
  Month 9: Usual activities (Moderate problem): number analyzed (Participants) | 10
  Month 9: Usual activities (Moderate problem) | 0
  Month 9: Usual activities (Severe problem): number analyzed (Participants) | 10
  Month 9: Usual activities (Severe problem) | 0
  Month 9: Usual activities (Unable to do usual activities): number analyzed (Participants) | 10
  Month 9: Usual activities (Unable to do usual activities) | 1
  Month 12: Usual activities (No problem): number analyzed (Participants) | 14
  Month 12: Usual activities (No problem) | 11
  Month 12: Usual activities (Slight problem): number analyzed (Participants) | 14
  Month 12: Usual activities (Slight problem) | 3
  Month 12: Usual activities (Moderate problem): number analyzed (Participants) | 14
  Month 12: Usual activities (Moderate problem) | 0
  Month 12: Usual activities (Severe problem): number analyzed (Participants) | 14
  Month 12: Usual activities (Severe problem) | 0
  Month 12: Usual activities (Unable to do usual activities): number analyzed (Participants) | 14
  Month 12: Usual activities (Unable to do usual activities) | 0
  Month 15: Usual activities (No problem): number analyzed (Participants) | 10
  Month 15: Usual activities (No problem) | 8
  Month 15: Usual activities (Slight problem): number analyzed (Participants) | 10
  Month 15: Usual activities (Slight problem) | 2
  Month 15: Usual activities (Moderate problem): number analyzed (Participants) | 10
  Month 15: Usual activities (Moderate problem) | 0
  Month 15: Usual activities (Severe problem): number analyzed (Participants) | 10
  Month 15: Usual activities (Severe problem) | 0
  Month 15: Usual activities (Unable to do usual activities): number analyzed (Participants) | 10
  Month 15: Usual activities (Unable to do usual activities) | 0
  Month 18: Usual activities (No problem): number analyzed (Participants) | 4
  Month 18: Usual activities (No problem) | 1
  Month 18: Usual activities (Slight problem): number analyzed (Participants) | 4
  Month 18: Usual activities (Slight problem) | 3
  Month 18: Usual activities (Moderate problem): number analyzed (Participants) | 4
  Month 18: Usual activities (Moderate problem) | 0
  Month 18: Usual activities (Severe problem): number analyzed (Participants) | 4
  Month 18: Usual activities (Severe problem) | 0
  Month 18: Usual activities (Unable to do usual activities): number analyzed (Participants) | 4
  Month 18: Usual activities (Unable to do usual activities) | 0
  Month 24: Usual activities (No problem): number analyzed (Participants) | 4
  Month 24: Usual activities (No problem) | 4
  Month 24: Usual activities (Slight problem): number analyzed (Participants) | 4
  Month 24: Usual activities (Slight problem) | 0
  Month 24: Usual activities (Moderate problem): number analyzed (Participants) | 4
  Month 24: Usual activities (Moderate problem) | 0
  Month 24: Usual activities (Severe problem): number analyzed (Participants) | 4
  Month 24: Usual activities (Severe problem) | 0
  Month 24: Usual activities (Unable to do usual activities): number analyzed (Participants) | 4
  Month 24: Usual activities (Unable to do usual activities) | 0
  Baseline: Pain/Discomfort (No Problem) | 23
  Baseline: Pain/Discomfort (Slight Problem) | 16
  Baseline: Pain/Discomfort (Moderate Problem) | 12
  Baseline: Pain/Discomfort (Severe Problem) | 0
  Baseline: Pain/Discomfort (Extreme Pain or discomfort) | 0
  Day 28: Pain/Discomfort (No Problem): number analyzed (Participants) | 42
  Day 28: Pain/Discomfort (No Problem) | 19
  Day 28: Pain/Discomfort (Slight Problem): number analyzed (Participants) | 42
  Day 28: Pain/Discomfort (Slight Problem) | 14
  Day 28: Pain/Discomfort (Moderate Problem): number analyzed (Participants) | 42
  Day 28: Pain/Discomfort (Moderate Problem) | 9
  Day 28: Pain/Discomfort (Severe Problem): number analyzed (Participants) | 42
  Day 28: Pain/Discomfort (Severe Problem) | 0
  Day 28: Pain/Discomfort (Extreme Pain or discomfort): number analyzed (Participants) | 42
  Day 28: Pain/Discomfort (Extreme Pain or discomfort) | 0
  Month 3: Pain/Discomfort (No Problem): number analyzed (Participants) | 26
  Month 3: Pain/Discomfort (No Problem) | 11
  Month 3: Pain/Discomfort (Slight Problem): number analyzed (Participants) | 26
  Month 3: Pain/Discomfort (Slight Problem) | 9
  Month 3: Pain/Discomfort (Moderate Problem): number analyzed (Participants) | 26
  Month 3: Pain/Discomfort (Moderate Problem) | 6
  Month 3: Pain/Discomfort (Severe Problem): number analyzed (Participants) | 26
  Month 3: Pain/Discomfort (Severe Problem) | 0
  Month 3: Pain/Discomfort (Extreme Pain or discomfort): number analyzed (Participants) | 26
  Month 3: Pain/Discomfort (Extreme Pain or discomfort) | 0
  Month 6: Pain/Discomfort (No Problem): number analyzed (Participants) | 25
  Month 6: Pain/Discomfort (No Problem) | 11
  Month 6: Pain/Discomfort (Slight Problem): number analyzed (Participants) | 25
  Month 6: Pain/Discomfort (Slight Problem) | 5
  Month 6: Pain/Discomfort (Moderate Problem): number analyzed (Participants) | 25
  Month 6: Pain/Discomfort (Moderate Problem) | 7
  Month 6: Pain/Discomfort (Severe Problem): number analyzed (Participants) | 25
  Month 6: Pain/Discomfort (Severe Problem) | 2
  Month 6: Pain/Discomfort (Extreme Pain or discomfort): number analyzed (Participants) | 25
  Month 6: Pain/Discomfort (Extreme Pain or discomfort) | 0
  Month 9: Pain/Discomfort (No Problem): number analyzed (Participants) | 10
  Month 9: Pain/Discomfort (No Problem) | 7
  Month 9: Pain/Discomfort (Slight Problem): number analyzed (Participants) | 10
  Month 9: Pain/Discomfort (Slight Problem) | 1
  Month 9: Pain/Discomfort (Moderate Problem): number analyzed (Participants) | 10
  Month 9: Pain/Discomfort (Moderate Problem) | 2
  Month 9: Pain/Discomfort (Severe Problem): number analyzed (Participants) | 10
  Month 9: Pain/Discomfort (Severe Problem) | 0
  Month 9: Pain/Discomfort (Extreme Pain or discomfort): number analyzed (Participants) | 10
  Month 9: Pain/Discomfort (Extreme Pain or discomfort) | 0
  Month 12: Pain/Discomfort (No Problem): number analyzed (Participants) | 14
  Month 12: Pain/Discomfort (No Problem) | 7
  Month 12: Pain/Discomfort (Slight Problem): number analyzed (Participants) | 14
  Month 12: Pain/Discomfort (Slight Problem) | 6
  Month 12: Pain/Discomfort (Moderate Problem): number analyzed (Participants) | 14
  Month 12: Pain/Discomfort (Moderate Problem) | 1
  Month 12: Pain/Discomfort (Severe Problem): number analyzed (Participants) | 14
  Month 12: Pain/Discomfort (Severe Problem) | 0
  Month 12: Pain/Discomfort (Extreme Pain or discomfort): number analyzed (Participants) | 14
  Month 12: Pain/Discomfort (Extreme Pain or discomfort) | 0
  Month 15: Pain/Discomfort (No Problem): number analyzed (Participants) | 10
  Month 15: Pain/Discomfort (No Problem) | 6
  Month 15: Pain/Discomfort (Slight Problem): number analyzed (Participants) | 10
  Month 15: Pain/Discomfort (Slight Problem) | 4
  Month 15: Pain/Discomfort (Moderate Problem): number analyzed (Participants) | 10
  Month 15: Pain/Discomfort (Moderate Problem) | 0
  Month 15: Pain/Discomfort (Severe Problem): number analyzed (Participants) | 10
  Month 15: Pain/Discomfort (Severe Problem) | 0
  Month 15: Pain/Discomfort (Extreme Pain or discomfort): number analyzed (Participants) | 10
  Month 15: Pain/Discomfort (Extreme Pain or discomfort) | 0
  Month 18: Pain/Discomfort (No Problem): number analyzed (Participants) | 4
  Month 18: Pain/Discomfort (No Problem) | 1
  Month 18: Pain/Discomfort (Slight Problem): number analyzed (Participants) | 4
  Month 18: Pain/Discomfort (Slight Problem) | 3
  Month 18: Pain/Discomfort (Moderate Problem): number analyzed (Participants) | 4
  Month 18: Pain/Discomfort (Moderate Problem) | 0
  Month 18: Pain/Discomfort (Severe Problem): number analyzed (Participants) | 4
  Month 18: Pain/Discomfort (Severe Problem) | 0
  Month 18: Pain/Discomfort (Extreme Pain or discomfort): number analyzed (Participants) | 4
  Month 18: Pain/Discomfort (Extreme Pain or discomfort) | 0
  Month 24: Pain/Discomfort (No Problem): number analyzed (Participants) | 4
  Month 24: Pain/Discomfort (No Problem) | 3
  Month 24: Pain/Discomfort (Slight Problem): number analyzed (Participants) | 4
  Month 24: Pain/Discomfort (Slight Problem) | 1
  Month 24: Pain/Discomfort (Moderate Problem): number analyzed (Participants) | 4
  Month 24: Pain/Discomfort (Moderate Problem) | 0
  Month 24: Pain/Discomfort (Severe Problem): number analyzed (Participants) | 4
  Month 24: Pain/Discomfort (Severe Problem) | 0
  Month 24: Pain/Discomfort (Extreme Pain or discomfort): number analyzed (Participants) | 4
  Month 24: Pain/Discomfort (Extreme Pain or discomfort) | 0
  Baseline: Anxiety/Depression (No problem) | 30
  Baseline: Anxiety/Depression (Slight problem) | 12
  Baseline: Anxiety/Depression (Moderate problem) | 7
  Baseline: Anxiety/Depression (Severe problem) | 2
  Baseline: Anxiety/Depression (Extreme Anxious or Depressed) | 0
  Day 28: Anxiety/Depression (No problem): number analyzed (Participants) | 42
  Day 28: Anxiety/Depression (No problem) | 28
  Day 28: Anxiety/Depression (Slight problem): number analyzed (Participants) | 42
  Day 28: Anxiety/Depression (Slight problem) | 11
  Day 28: Anxiety/Depression (Moderate problem): number analyzed (Participants) | 42
  Day 28: Anxiety/Depression (Moderate problem) | 3
  Day 28: Anxiety/Depression (Severe problem): number analyzed (Participants) | 42
  Day 28: Anxiety/Depression (Severe problem) | 0
  Day 28: Anxiety/Depression (Extreme Anxious or Depressed): number analyzed (Participants) | 42
  Day 28: Anxiety/Depression (Extreme Anxious or Depressed) | 0
  Month 3: Anxiety/Depression (No problem): number analyzed (Participants) | 26
  Month 3: Anxiety/Depression (No problem) | 17
  Month 3: Anxiety/Depression (Slight problem): number analyzed (Participants) | 26
  Month 3: Anxiety/Depression (Slight problem) | 6
  Month 3: Anxiety/Depression (Moderate problem): number analyzed (Participants) | 26
  Month 3: Anxiety/Depression (Moderate problem) | 3
  Month 3: Anxiety/Depression (Severe problem): number analyzed (Participants) | 26
  Month 3: Anxiety/Depression (Severe problem) | 0
  Month 3: Anxiety/Depression (Extreme Anxious or Depressed): number analyzed (Participants) | 26
  Month 3: Anxiety/Depression (Extreme Anxious or Depressed) | 0
  Month 6: Anxiety/Depression (No problem): number analyzed (Participants) | 25
  Month 6: Anxiety/Depression (No problem) | 18
  Month 6: Anxiety/Depression (Slight problem): number analyzed (Participants) | 25
  Month 6: Anxiety/Depression (Slight problem) | 4
  Month 6: Anxiety/Depression (Moderate problem): number analyzed (Participants) | 25
  Month 6: Anxiety/Depression (Moderate problem) | 3
  Month 6: Anxiety/Depression (Severe problem): number analyzed (Participants) | 25
  Month 6: Anxiety/Depression (Severe problem) | 0
  Month 6: Anxiety/Depression (Extreme Anxious or Depressed): number analyzed (Participants) | 25
  Month 6: Anxiety/Depression (Extreme Anxious or Depressed) | 0
  Month 9: Anxiety/Depression (No problem): number analyzed (Participants) | 10
  Month 9: Anxiety/Depression (No problem) | 9
  Month 9: Anxiety/Depression (Slight problem): number analyzed (Participants) | 10
  Month 9: Anxiety/Depression (Slight problem) | 0
  Month 9: Anxiety/Depression (Moderate problem): number analyzed (Participants) | 10
  Month 9: Anxiety/Depression (Moderate problem) | 1
  Month 9: Anxiety/Depression (Severe problem): number analyzed (Participants) | 10
  Month 9: Anxiety/Depression (Severe problem) | 0
  Month 9: Anxiety/Depression (Extreme Anxious or Depressed): number analyzed (Participants) | 10
  Month 9: Anxiety/Depression (Extreme Anxious or Depressed) | 0
  Month 12: Anxiety/Depression (No problem): number analyzed (Participants) | 14
  Month 12: Anxiety/Depression (No problem) | 10
  Month 12: Anxiety/Depression (Slight problem): number analyzed (Participants) | 14
  Month 12: Anxiety/Depression (Slight problem) | 2
  Month 12: Anxiety/Depression (Moderate problem): number analyzed (Participants) | 14
  Month 12: Anxiety/Depression (Moderate problem) | 2
  Month 12: Anxiety/Depression (Severe problem): number analyzed (Participants) | 14
  Month 12: Anxiety/Depression (Severe problem) | 0
  Month 12: Anxiety/Depression (Extreme Anxious or Depressed): number analyzed (Participants) | 14
  Month 12: Anxiety/Depression (Extreme Anxious or Depressed) | 0
  Month 15: Anxiety/Depression (No problem): number analyzed (Participants) | 10
  Month 15: Anxiety/Depression (No problem) | 7
  Month 15: Anxiety/Depression (Slight problem): number analyzed (Participants) | 10
  Month 15: Anxiety/Depression (Slight problem) | 2
  Month 15: Anxiety/Depression (Moderate problem): number analyzed (Participants) | 10
  Month 15: Anxiety/Depression (Moderate problem) | 1
  Month 15: Anxiety/Depression (Severe problem): number analyzed (Participants) | 10
  Month 15: Anxiety/Depression (Severe problem) | 0
  Month 15: Anxiety/Depression (Extreme Anxious or Depressed): number analyzed (Participants) | 10
  Month 15: Anxiety/Depression (Extreme Anxious or Depressed) | 0
  Month 18: Anxiety/Depression (No problem): number analyzed (Participants) | 4
  Month 18: Anxiety/Depression (No problem) | 3
  Month 18: Anxiety/Depression (Slight problem): number analyzed (Participants) | 4
  Month 18: Anxiety/Depression (Slight problem) | 1
  Month 18: Anxiety/Depression (Moderate problem): number analyzed (Participants) | 4
  Month 18: Anxiety/Depression (Moderate problem) | 0
  Month 18: Anxiety/Depression (Severe problem): number analyzed (Participants) | 4
  Month 18: Anxiety/Depression (Severe problem) | 0
  Month 18: Anxiety/Depression (Extreme Anxious or Depressed): number analyzed (Participants) | 4
  Month 18: Anxiety/Depression (Extreme Anxious or Depressed) | 0
  Month 24: Anxiety/Depression (No problem): number analyzed (Participants) | 4
  Month 24: Anxiety/Depression (No problem) | 4
  Month 24: Anxiety/Depression (Slight problem): number analyzed (Participants) | 4
  Month 24: Anxiety/Depression (Slight problem) | 0
  Month 24: Anxiety/Depression (Moderate problem): number analyzed (Participants) | 4
  Month 24: Anxiety/Depression (Moderate problem) | 0
  Month 24: Anxiety/Depression (Severe problem): number analyzed (Participants) | 4
  Month 24: Anxiety/Depression (Severe problem) | 0
  Month 24: Anxiety/Depression (Extreme Anxious or Depressed): number analyzed (Participants) | 4
  Month 24: Anxiety/Depression (Extreme Anxious or Depressed) | 0

18. Secondary Outcome: Phase 2: EQ-5D Visual Analogue Scale (VAS) Score
Description: EQ-5D is a self-reported questionnaire used for assessing the overall health status of a participant. The EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single index value. The EQ-5D-VAS records the participant's self-rated health on a 20-cm vertical visual analogue scale and is asked to make a global assessment of their current state of health with 0 indicating the worst health they can imagine and 100 indicating the best health they can imagine. Higher scores indicated a better health state.
Time Frame: Baseline, Day 28, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, and Month 24
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
Number analyzed (Participants) | 51
score on a scale
  Baseline | 68.2 (21.8)
  Day 28: number analyzed (Participants) | 41
  Day 28 | 74.7 (17.9)
  Month 3: number analyzed (Participants) | 26
  Month 3 | 79.7 (12.2)
  Month 6: number analyzed (Participants) | 25
  Month 6 | 81.0 (17.6)
  Month 9: number analyzed (Participants) | 10
  Month 9 | 81.7 (23.1)
  Month 12: number analyzed (Participants) | 14
  Month 12 | 86.9 (10.0)
  Month 15: number analyzed (Participants) | 10
  Month 15 | 87.8 (11.6)
  Month 18: number analyzed (Participants) | 4
  Month 18 | 93.3 (5.9)
  Month 24: number analyzed (Participants) | 4
  Month 24 | 97.5 (2.9)

ADVERSE EVENTS:
Time Frame: Adverse Event: Up to 5 years; All-Cause mortality: Up to to 7.1 years
Description: Adverse Events: The Safety Analysis Set included all participants treated with any dose of brexucabtagene autoleucel.
  All-cause mortality: All Enrolled Analysis Set included all enrolled participants in the study.
Arm/Group | Phase 1: 2 x 10^6 Anti-CD19 CAR T Cells/kg | Phase 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg | Phase 1: 0.5 x 10^6 Anti-CD19 CAR T Cells/kg | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg
All-Cause Mortality (participants affected / at risk) | 6/6 | 17/28 | 15/20 | 39/71
Serious Adverse Events (participants affected / at risk) | 6/6 | 21/23 | 12/16 | 41/55
Other Adverse Events (participants affected / at risk) | 6/6 | 23/23 | 16/16 | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 2 x 10^6 Anti-CD19 CAR T Cells/kg (N=6) | Phase 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg (N=23) | Phase 1: 0.5 x 10^6 Anti-CD19 CAR T Cells/kg (N=16) | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg (N=55)
Cytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 4 | 1 | 15
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Graft versus host disease (Immune system disorders) | 0 | 1 | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 2
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Device related bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 2 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes simplex viraemia (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis fungal (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 3
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 4 | 3 | 2
Septic shock (Infections and infestations) | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 4 | 4
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 3 | 1 | 3
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 2 | 8 | 1 | 4
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 2
Seizure (Nervous system disorders) | 0 | 1 | 1 | 3
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 3
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 9 | 3 | 16
Shock (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 2 x 10^6 Anti-CD19 CAR T Cells/kg (N=6) | Phase 1: 1 x 10^6 Anti-CD19 CAR T Cells/kg (N=23) | Phase 1: 0.5 x 10^6 Anti-CD19 CAR T Cells/kg (N=16) | Phase 2: 1 x 10^6 Anti-CD19 CAR T Cells/kg (N=55)
Anaemia (Blood and lymphatic system disorders) | 3 | 14 | 4 | 29
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Bone marrow reticulin fibrosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 2 | 5
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 7 | 1 | 8
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 9
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 2 | 5
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 4 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 2 | 8 | 2 | 19
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 4 | 6 | 13
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 3
Eye pain (Eye disorders) | 0 | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 1 | 2
Vision blurred (Eye disorders) | 0 | 3 | 2 | 4
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 5 | 2 | 10
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 11 | 2 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 11 | 6 | 11
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Ileus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 11 | 3 | 21
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 7 | 2 | 9
Asthenia (General disorders) | 0 | 3 | 1 | 3
Catheter site pain (General disorders) | 1 | 0 | 0 | 1
Chills (General disorders) | 3 | 12 | 3 | 18
Face oedema (General disorders) | 0 | 0 | 1 | 3
Fatigue (General disorders) | 1 | 7 | 6 | 13
Gravitational oedema (General disorders) | 1 | 0 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 5
Non-cardiac chest pain (General disorders) | 0 | 2 | 1 | 2
Oedema (General disorders) | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 1 | 7 | 4 | 10
Pain (General disorders) | 0 | 3 | 0 | 7
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 6 | 21 | 11 | 49
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 0 | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 1 | 3 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 3 | 0 | 3
Bacteraemia (Infections and infestations) | 1 | 1 | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 3
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 8 | 0 | 12
Aspartate aminotransferase increased (Investigations) | 1 | 9 | 0 | 10
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 4
Blood bilirubin increased (Investigations) | 2 | 4 | 0 | 3
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 2
Blood fibrinogen decreased (Investigations) | 0 | 4 | 0 | 2
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 4
Neutrophil count decreased (Investigations) | 0 | 8 | 4 | 15
Platelet count decreased (Investigations) | 1 | 10 | 5 | 18
Weight decreased (Investigations) | 3 | 3 | 0 | 1
Weight increased (Investigations) | 2 | 2 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 2 | 4 | 14
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 9 | 4 | 8
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 8 | 5 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 5 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 8 | 1 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 11 | 2 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 8 | 1 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 7 | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 13 | 3 | 15
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 2
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 3
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0 | 6
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2
Aphasia (Nervous system disorders) | 0 | 8 | 3 | 6
Ataxia (Nervous system disorders) | 0 | 2 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 3
Dizziness (Nervous system disorders) | 1 | 2 | 2 | 8
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 4 | 6 | 1 | 9
Headache (Nervous system disorders) | 1 | 10 | 8 | 20
Lethargy (Nervous system disorders) | 0 | 3 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 1 | 3
Tremor (Nervous system disorders) | 1 | 8 | 4 | 15
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 4 | 2 | 7
Anxiety (Psychiatric disorders) | 1 | 5 | 2 | 4
Confusional state (Psychiatric disorders) | 2 | 6 | 6 | 11
Delirium (Psychiatric disorders) | 2 | 0 | 2 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 3 | 0 | 7
Mental status changes (Psychiatric disorders) | 0 | 2 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 2 | 3
Urinary retention (Renal and urinary disorders) | 1 | 3 | 2 | 2
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 5 | 12
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 2
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 3
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 2 | 5
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Distributive shock (Vascular disorders) | 0 | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 3 | 1 | 3
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 3 | 2 | 7
Hypotension (Vascular disorders) | 5 | 13 | 7 | 27
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
CRS (Immune system disorders) | 6 | 23 | 13 | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol: Amendment 6 (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT02614066/Prot_000.pdf
  • Study Protocol: Amendment 7 (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT02614066/Prot_002.pdf
  • Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT02614066/SAP_001.pdf